CLINICAL TRIAL: NCT03553238
Title: An Open-Label, One-Arm, Multi-Site Trial of Precision Diagnosis Directing Histone Deacetylase Inhibitor Chidamide Target Total Therapy for Adult Early T-cell Progenitor Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Precision Diagnosis Directing HDACi Chidamide Target Therapy for Adult ETP-ALL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, M.D., Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT-ETP-ALL
Record Dates: First submitted 2018-04-21; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Leukemia, Acute; Leukemia, T Cell; Leukemia, Lymphoblastic
Keywords: Early T-cell Precursor; Acute Lymphoblastic Leukemia; Histone Deacetylase Inhibitor; Chidamide
MeSH Terms: conditions — Leukemia; Leukemia, T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Dexamethasone; Vincristine; Cyclophosphamide; Idarubicin; pegaspargase; Doxorubicin; Methotrexate; Mercaptopurine; Etoposide; Cytarabine; Injections, Spinal; Radiotherapy; Karyotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETP-ALL (Experimental): Chidamide at a dose of 10mg/day will be added to PDT-ETP-ALL protocol. The intervention of PDT-ETP-ALL consists of diagnostic test (bone marrow aspiration, flow immunophenotyping, Karyotyping ，FISH, NGS, Flow-MRD, PET-CT scan), induction regimen (chidamide, dexamethasone, vincristine, cyclophosphamide, idarubicin, pegaspargase), consolidation regimen (chidamide, prednisone, cytarabine, methotrexate, cyclophosphamide, etoposide, adriamycin, 6-mercaptopurine, pegaspargase), MRD assessment and maintenance regimen (chidamide, prednisone, vincristine, methotrexate, 6-mercaptopurine), intrathecal injection chemotherapy, radiation therapy (for mediastinum- and/or central nervous system-involved lymphoma/leukemia) and allogeneic hematopoietic stem cell transplantation for patients with donor.
  Interventions: Drug: Chidamide; Drug: Dexamethasone; Drug: vincristine; Drug: Cyclophosphamide; Drug: Idarubicin; Drug: Pegaspargase; Drug: Adriamycin; Drug: Methotrexate; Drug: 6-Mercaptopurine; Drug: Etoposide; Drug: Cytarabine; Procedure: Bone marrow aspiration; Procedure: Intrathecal injection; Radiation: Radiation therapy; Genetic: NGS; Procedure: allogeneic hematopoietic stem cell transplantation; Diagnostic Test: Flow-MRD; Diagnostic Test: FISH; Diagnostic Test: Flow immunophenotyping; Diagnostic Test: Karyotyping

INTERVENTIONS:
Drug: Chidamide — Chidamide will be administrated at a dose of 10mg/day in PDT-ETP-ALL protocol.
  Other Names: HDACi chidamide
Drug: Dexamethasone — Dexamethasone will be added in Pre-phase Regimen, Induction-Regimen, Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: DXM
Drug: vincristine — Vincristine will be added to Induction-Regimen, Consolidation-Module and Maintenance-Module of PDT-ETP-ALL protocol.
  Other Names: VCR
Drug: Cyclophosphamide — CTX will be added to Induction-Regimen, Consolidation-Module and Maintenance-Module of PDT-ETP-ALL protocol.
  Other Names: CTX
Drug: Idarubicin — IDA will be added to Induction-Regimen and Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: IDA
Drug: Pegaspargase — PEG-ASP will be added to Induction-Regimen and Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: PEG-ASP
Drug: Adriamycin — Adriamycin will be added to Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: ADR
Drug: Methotrexate — Methotrexate will be added to consolidation module of PDT-ETP-ALL protocol.
  Other Names: MTX
Drug: 6-Mercaptopurine — Mercaptopurine will be added to Consolidation-Module and Maintenance-Module of PDT-ETP-ALL protocol.
  Other Names: 6-MP
Drug: Etoposide — VP-16 will be added to Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: VP-16
Drug: Cytarabine — AraC will be added to Consolidation-Module of PDT-ETP-ALL protocol.
  Other Names: AraC
Procedure: Bone marrow aspiration — Bone marrow aspiration and additional tests will be performed in all module of PDT-ETP-ALL protocol.
  Other Names: BM test
Procedure: Intrathecal injection — Intrathecal injection chemotherapy will be performed in PDT-ETP-ALL protocol.
  Other Names: IT
Radiation: Radiation therapy — Radiation therapy will be performed for mediastinum and/or central nervous system leukemia in PDT-ETP-ALL protocol.
  Other Names: RT
Genetic: NGS — Next-Generation-Sequencing (NGS) will be performed in PDT-ETP-ALL protocol.
Procedure: allogeneic hematopoietic stem cell transplantation — Allo-HSCT will be performed for patients with available donor in PDT-ETP-ALL protocol.
  Other Names: allo-HSCT
Diagnostic Test: Flow-MRD — Flow-MRD will be added to PDT-ETP-ALL for bone marrow and cerebrospinal fluid samples.
Diagnostic Test: FISH — FISH will be performed in PDT-ETP-ALL for bone marrow samples.
Diagnostic Test: Flow immunophenotyping — Flow immunophenotyping will be performed in PDT-ETP-ALL protocol.
Diagnostic Test: Karyotyping — Karyotyping will be performed in PDT-ETP-ALL protocol.

SUMMARY:
ETP-ALL is a recently recognized high-risk subgroup and the optimal therapeutic approaches are poorly characterized. Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, one-arm, multi-site trial is aimed to evaluate the safety and effect of a novel oral histone deacetylase inhibitor chidamide for adult ETP-ALL/LBL in CHINA.

DETAILED DESCRIPTION:
Early T-cell precursor (ETP) lymphoblastic leukemia (ETP-ALL) is a neoplasm composed of cells committed to the T-cell lineage but with an unique immunophenotype indicating only limited early T differentiation. In the highly orchestrated development of T cell fate specification under physiological condition, the most immature early thymic progenitors (ETPs) retain multilineage potentials. ETP-ALL blasts have a characteristic immunophenotype, with reduced/absent expression of T-lymphoid markers CD1a, CD5, CD8; and positivity for at least one HSC and/or myeloid antigen CD34, CD117, HLA-DR, CD13, CD33, CD11b, CD65. Recent study shed light on the genetic landscape of adult ETP-ALL, which revealed that more than 40% adult ETP-ALL harbored histone modification mutations. Chidamide is a novel oral HDACi with promising activity in non-Hodgkin lymphoma (NHL). Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, one-arm, multi-site trial is aimed to evaluate the safety and effect of a novel oral histone deacetylase inhibitor chidamide for adult ETP-ALL/LBL. HDACi chidamide at a dose of 10mg/day will be added to ETP-ALL group from induction therapy to consolidation therapy (total courses of chidamide treatment: 5 courses for allo-HSCT after Consolidation Module-3; 12 courses for patients non-allo-HSCT after Consolidation Module 1-9). Primary study endpoint of PDT-ETP-ALL is event-free survival of ETP-ALL group and secondary study endpoints are complete remission and MRD after induction, adverse event and overall survival of ETP-ALL group.

Pretreatment: Dexamethasone, -3 to 0d;

Induction:VCR: 1, 8, 15, 22; IDA: 1, 8; CTX: 1g/m2, 1, 8; PEG-asp: 2000-2500IU/m2, 1, 15; Dex: 1-24, chidamide: 10mg/d, po, qd.

MRD: d14, 24, 45, and pre-allo-HSCT.

VLCAM (MRD1/d14>1%): CTX, d25; AraC 2g/m2, q12h, d25, 26; 6-MP: 25-31, PEG-asp: 26; chidamide: 10mg/d, po, qd.

Consolidation Module:

CM-1: AraC 3g/m2, q12h, 1-2, Dex: 10mg/m2, 1-2, PEG-asp: 2, 6-MP: 1-7. IT: d1, chidamide: 10mg/d, po, qd.

CM-2: MTX 5g/m2, 1, Dex: 10mg/m2, 1-2, PEG-asp: 2; 6-MP: 1-7; IT: d1; chidamide: 10mg/d, po, qd.

CM-3: CTX 0.5g/m2, 1-3, PEG-asp: 2, Doxorubicin: 40mg/m2, 4, 6-MP: 1-7, IT: d1;chidamide: 10mg/d, po, qd.

Allo-HSCT: after CM-3 when donors available. Non-HSCT: finish CM 4-9 and POMP maintenance.

CM 4-6: repeat CM 1-3. Re-Induction: after CM-6. CM 7-9: repeat CM1-3.

Maintenance: CPOMP-chidamide 10mg/d, po, qd; Pred for 12 months; VCR for 12 months; MTX for 24 months; 6-MP for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 14-55 years old;
* ETP-ALL newly diagnosed;
* signed written informed consent

Exclusion Criteria:

* Pregnant women;
* History of pancreatitis;
* History of diabetes;
* History of active peptic ulcer disease in the past 6 months;
* History of arteriovenous thrombosis in the past 6 months;
* Severe active infection;
* Allergic to any drugs in PDT-ETP-ALL.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02-14 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years

SECONDARY OUTCOMES:
Minimum residual disease after induction | 3 months
CR after Induction Therapy | 3 years
Death in induction | 3 month
Adverse events | 3 years
Relapse | 3 years
Relapse free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Zhou, MD, PhD, Study Director — Nanfang Hospital, Southern Medical University, CHINA
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Koch U, Radtke F. Mechanisms of T cell development and transformation. Annu Rev Cell Dev Biol. 2011;27:539-62. doi: 10.1146/annurev-cellbio-092910-154008. Epub 2011 Jul 5. PMID 21740230
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Bond J, Graux C, Lhermitte L, Lara D, Cluzeau T, Leguay T, Cieslak A, Trinquand A, Pastoret C, Belhocine M, Spicuglia S, Lheritier V, Lepretre S, Thomas X, Huguet F, Ifrah N, Dombret H, Macintyre E, Boissel N, Asnafi V. Early Response-Based Therapy Stratification Improves Survival in Adult Early Thymic Precursor Acute Lymphoblastic Leukemia: A Group for Research on Adult Acute Lymphoblastic Leukemia Study. J Clin Oncol. 2017 Aug 10;35(23):2683-2691. doi: 10.1200/JCO.2016.71.8585. Epub 2017 Jun 12. PMID 28605290
- [Background] Yu S, Zhou X, Steinke FC, Liu C, Chen SC, Zagorodna O, Jing X, Yokota Y, Meyerholz DK, Mullighan CG, Knudson CM, Zhao DM, Xue HH. The TCF-1 and LEF-1 transcription factors have cooperative and opposing roles in T cell development and malignancy. Immunity. 2012 Nov 16;37(5):813-26. doi: 10.1016/j.immuni.2012.08.009. Epub 2012 Oct 25. PMID 23103132
- [Derived] Lin J, Huang Z, Cai Z, Li J, Li Z, Ding C, Wang Z, Li X, Zhou X, He B, Zhong W, Xuan L, Liu Q, Xu Y, Zhou H. Tucidinostat plus pediatric-inspired chemotherapy for newly diagnosed adult ETP-ALL/LBL: a single-arm, phase 2 trial. J Hematol Oncol. 2024 Oct 28;17(1):101. doi: 10.1186/s13045-024-01624-8. PMID 39468701